CLINICAL TRIAL: NCT07186010
Title: Immunogenomic Dynamics and Biomarkers in Patients With Hepatocellular Carcinoma Receiving Immunotherapy
Status: Recruiting | Type: Observational
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Ju Hyun Shim, Professor, Asan Medical Center
Other Study IDs: KCT0005305
Record Dates: First submitted 2025-09-08; First posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Hepatocellular Carcinoma; Liver Cancer
Keywords: immunotherapy; biomarker; HCC
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — blood samples containing circulating tumor DNA
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
1. Research purpose To perform genomic and immune profiling analysis on blood and tissue samples obtained from blood sampling and tumor biopsy in patients with advanced hepatocellular carcinoma with immuno-oncology treatment.
2. Research Subject Patients who will receive immuno-oncology treatment in recurrent, metastatic, and advanced liver cancer, who meet the selection criteria of the study, do not have exclusion criteria, and voluntarily agree to participate in the study.
3. Number of study subjects 50 people
4. Research Method 1) In patients with advanced hepatocellular carcinoma, peripheral blood will be collected at baseline before treatment, 6 weeks, 12 weeks, 24 weeks, 48 weeks after treatment, and at the time of cancer progression.

2) Fresh tumors will be stored in the tissue obtained during the biopsy to perform genetic analysis

DETAILED DESCRIPTION:
This study is designed to perform comprehensive genomic and immune profiling in patients with advanced hepatocellular carcinoma (HCC) undergoing immuno-oncology (IO) treatment. The objective is to investigate molecular and immunologic biomarkers in both blood and tumor tissue that may correlate with treatment response, disease progression, and clinical outcomes.

Eligible patients include those with recurrent, metastatic, or advanced HCC who are scheduled to receive IO therapy and who meet the study's inclusion and exclusion criteria. Approximately 50 participants will be enrolled.

Peripheral blood samples will be collected at predefined time points: prior to initiation of IO treatment (baseline), and at 6, 12, 24, and 48 weeks after treatment initiation, as well as at the time of disease progression. These blood samples will be subjected to genomic and immune profiling, including but not limited to circulating tumor DNA analysis, immune cell subset characterization, and cytokine/chemokine profiling.

In addition, fresh tumor tissue obtained from biopsy procedures will be stored and used for genetic and immunologic analyses. Tissue-based studies may include next-generation sequencing, immunohistochemistry, multiplex immunofluorescence, and other exploratory assays to evaluate tumor mutational landscape, immune checkpoint expression, and tumor microenvironmental features.

By integrating longitudinal blood-based biomarkers with tumor tissue data, this study aims to better characterize tumor biology, immune dynamics, and mechanisms of resistance in advanced HCC treated with immuno-oncology agents. The ultimate goal is to identify predictive and prognostic biomarkers that may guide personalized treatment strategies and improve clinical outcomes in this patient population.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically confirmed HCC,
2. Patients with histologically confirmed locally advanced, recurrent or metastatic HCC, which was judged not to be eligible for surgical resection, liver transplantation or radiofrequency ablation
3. Patients who will receive immuno-oncology treatment

Exclusion Criteria:

1. Patients with histologically confirmed fibrolamellar type HCC, sarcomatoid HCC, or mixed cholangiocarcinoma and HCC
2. Patients with concurrent other malignancy
3. Patients who are candidates for local curative treatments such as hepatic resection, liver transplantation, or radiofrequency ablation
4. Patients who have a possibility of confusion in the results of the clinical research

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with histologically confirmed recurrent, locally advanced or metastatic HCC who will receive immuno-oncology treatment
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-09-28 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) according to RECIST 1.1 criteria | from the date of the first immunotherapy date', every 9 weeks, for 2 years
  Proportion of participants achieving complete response (CR) or partial response (PR) as their best overall response, assessed by imaging according to RECIST 1.1 criteria.

SECONDARY OUTCOMES:
overall survival | From date of immunotherapy until the date of death from any cause or study end whichever came first, assessed up to assessed up to 5 years
  overall survival after initiation of immunotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Ju Hyun Shim, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, Song-pa, South Korea